CLINICAL TRIAL: NCT00472823
Title: Determination of RDA for Vitamin D in Caucasian and African American Women
Brief Title: Vitamin D Supplementation in Older Women
Acronym: VIDOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Creighton University (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Office of Dietary Supplements (ODS) (NIH); University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AG0081; 1R01AG028168-01 (NIH)
Record Dates: First submitted 2007-05-10; First posted 2007-05-14 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-03

CONDITIONS: Osteoporosis; Aging
Keywords: cholecalciferol; vitamin D deficiency; bone density; dietary calcium; hypercalcemia; hypercalciuria
MeSH Terms: conditions — Osteoporosis; Vitamin D Deficiency; Hypercalcemia; Hypercalciuria | interventions — Cholecalciferol; Calcium Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- vitamin D3 400 IU daily (Experimental): vitamin D3 400 IU daily
  Interventions: Dietary Supplement: Vitamin D3; Dietary Supplement: Calcium Citrate (Citracal)
- vitamin D3 800 IU daily (Experimental): vitamin D3 800 IU daily
  Interventions: Dietary Supplement: Vitamin D3; Dietary Supplement: Calcium Citrate (Citracal)
- vitamin D3 1600 IU daily (Experimental): vitamin D3 1600 IU daily
  Interventions: Dietary Supplement: Vitamin D3; Dietary Supplement: Calcium Citrate (Citracal)
- vitamin D3 2400 IU daily (Experimental): vitamin D3 2400 IU daily
  Interventions: Dietary Supplement: Vitamin D3; Dietary Supplement: Calcium Citrate (Citracal)
- vitamin D3 3200 IU daily (Experimental): vitamin D3 3200 IU daily
  Interventions: Dietary Supplement: Vitamin D3; Dietary Supplement: Calcium Citrate (Citracal)
- vitamin D3 4000 IU daily (Experimental): vitamin D3 4000 IU daily
  Interventions: Dietary Supplement: Vitamin D3; Dietary Supplement: Calcium Citrate (Citracal)
- vitamin D3 4800 IU daily (Experimental): vitamin D3 4800 IU daily
  Interventions: Dietary Supplement: Vitamin D3; Dietary Supplement: Calcium Citrate (Citracal)
- placebo (Placebo Comparator): matched to vitamin D tablet
  Interventions: Dietary Supplement: Vitamin D3

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — Orally for one year
Dietary Supplement: Calcium Citrate (Citracal) — Orally for one year; dosage adjusted so that calcium intake is 1200-1400mg daily
  Other Names: Citracal
  Arms: vitamin D3 1600 IU daily; vitamin D3 2400 IU daily; vitamin D3 3200 IU daily; vitamin D3 400 IU daily; vitamin D3 4000 IU daily; vitamin D3 4800 IU daily; vitamin D3 800 IU daily

SUMMARY:
The purpose of this study is to examine the effects of several doses of vitamin D on hormones related to bone, calcium absorption, bone density and muscle strength.

DETAILED DESCRIPTION:
The prevalence of osteoporosis is high in the United States, with about 10 million people over the age of 50 already having the disease and another 34 million at risk for developing it. Development of low-cost and effective strategies is important for preventing osteoporosis and reducing osteoporotic fractures. A simple inexpensive strategy to prevent osteoporosis is adequate nutrition with calcium and vitamin D. Serum 25OHD (25-hydroxyvitamin D) is now accepted as the objective measure of vitamin D nutrition. There is a growing understanding that serum 25OHD concentrations of at least 30-32 ng/ml are needed for optimal bone health at which serum parathyroid hormone (PTH) concentrations reach a minimum.

There are no systematic prospective dose response studies aimed at determining the optimum amount of vitamin D intake required to maintain optimum serum 25OHD levels in the population which will help in determining the estimated average requirement (EAR) and recommended dietary requirement (RDA) for vitamin D. More work to determine the RDA for vitamin D has been recommended by the Panel on Calcium and Related Nutrients of the Food and Nutrition Board. This study is aimed at filling the information gap by concentrating on the high risk group of postmenopausal women. We are testing the theory that increasing serum 25OHD to a level greater than 30 ng/ml will reduce serum PTH in the high risk group of vitamin D insufficient postmenopausal women with an adequate intake of calcium. We also believe that the dose of vitamin D that will achieve this level is approximately 4400IU per day, which is well above the suggested adequate intake of 400-600 ID recommended for the elderly.

In a one year double blind, randomized prospective clinical trial, we will examine the dose response effect of supplementation with different doses of vitamin D3 (400, 800, 1600, 2400, 3200, 4000, 4800IU/day) on the primary outcomes of serum 25OHD and PTH in 160 postmenopausal Caucasian and 160 African American women who have inadequate vitamin D levels in winter. We expect that the results from this study will add useful and important information about the RDA for vitamin D for postmenopausal women who are more susceptible to osteoporosis. The results from this study will also help in designing future clinical trials to study the effect of vitamin D, for example in preventing fractures, falls, cancer.

The main objective of the current proposal is to study the effect of increasing doses of vitamin D3 in the high risk group of postmenopausal Caucasian and African American women with hypovitaminosis D (serum 25OHD <20 ng/ml) in winter in presence of sufficient calcium intake, in order to determine the Estimated Average Requirement (EAR) that covers 50% and the Recommended Daily allowance (RDA) covers 97.5% of population for vitamin D. We will use a serum 25OHD concentration equal >30 ng/ml and normalization of serum PTH as indicators of adequacy. We expect that the results from this proposal will add important information helpful in designing future larger clinical trials to determine the recommended dietary allowance (RDA) for vitamin D in other ethnic groups and designing clinical trials on the effect of vitamin D on falls and fractures.

We hypothesize that increasing serum 25OHD to a level greater than 30 ng/ml with vitamin D supplements in 97 percent of the study subjects will reduce serum PTH and bone markers to premenopausal range. We postulate that the RDA of vitamin D that will achieve a serum 25OHD of ≥ 30 ng/ml in 97.5% of women during winter is approximately 4400 IU/d and the EAR dose of vitamin D is between 800-1000 IU.

The specific aims of the proposal are,

1. To examine the dose response effect of vitamin D3, 400, 800, 1600, 2400, 3200, 4000, and 4800 IU /d in postmenopausal Caucasian and African American women with hypovitaminosis D (serum 25OHD equal <20 ng/ml) in winter plus an adequate calcium intake compared to a calcium control group, on serum 25OHD and PTH levels, which constitute our primary outcome measures.
2. To determine the EAR and RDA for postmenopausal women by establishing the dose of vitamin D3 that will increase serum 25OHD above 30 ng/ml in 97.5% of study subjects in winter and reduce serum PTH to the normal premenopausal range.
3. To study the dose response effect of vitamin D3 on calcium absorption, 1,25-dihydroxyvitamin D3 (1,25(OH)2D3) serum calcium, serum bone markers, bone mineral density (BMD) and falls (only in elderly) (the secondary outcome measures)
4. To establish the long term safety of these doses relating to hypercalcemia and hypercalciuria

Progress: Caucasian enrollment completed July 2008; African American enrollment completed May 2009

ELIGIBILITY:
Inclusion Criteria:

* At least 7 years post-menopause
* Serum 25OHD level 5 ng/ml to 20 ng/ml
* BMI less than or equal to 40 kg/m2
* Willing to discontinue multivitamins that contain vitamin D during the study

Exclusion Criteria:

* Cancer (except basal cell carcinoma) or terminal illness
* Previous hip fracture
* Hemiplegia (paralysis of one side of the body)
* Uncontrolled type I diabetes or fasting blood sugar greater than 140 mg in type II
* Kidney stones more than twice in a lifetime
* Chronic renal failure
* Evidence of chronic liver disease, including alcoholism
* Physical conditions such as severe osteoarthritis, rheumatoid arthritis, heart failure severe enough to prevent reasonable physical activity
* Previous treatment with bisphosphonates (more that 3 months), PTH or PTH derivatives, (e.g. Teriparatide or Fluoride) in the last 6 months
* Previous treatment within the last 6 months with calcitonin or estrogen
* Chronic high dose corticosteroid therapy (more than 10 mg per day) for over 6 months and not within the last 6 months
* Anticonvulsant therapy
* High dose thiazide therapy (more than 37.5 mg)
* 24 hour urine calcium greater than 290 mg on 2 baseline tests
* Serum calcium exceeding upper normal limit on 2 baseline tests
* Bone Mineral Density T-score less than -3.0 for spine or hip

Min Age: 57 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2007-04; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Changes in Serum 25-hydroxyvitamin D (25OHD) and parathyroid hormone (PTH) levels | Baseline, 6months,12 months

SECONDARY OUTCOMES:
Calcium absorption | Baseline and 12 months
  100mg calcium+ calcium45
Serum/urine calcium | Baseline and every 3 months
Bone markers | Baseline, and 12 months
Bone density | Baseline and 12 months
  spine,hip,total body,lateral
Muscle strength | Baseline,6 months,12 months
  leg strength( Cybex),timed up and go,hand grip,chair stand,gait speed,quiet stance,postural stability( biodex),standing balance
Falls | Baseline and every 3 months
  questionnaire
Pulmonary function studies | baseline and final test
  FEV1
Genotyping | one time
Molecular studies of peripheral leucocytes | baseline and final test
Adult Depression Score | baseline and 12 months
  questionnaire
Physical Activity Scale form ( PASE) | baseline,6 months,12 months
  questionnaire
sun exposure | baseline and every 3 months
  sun exposure form and skin color evaluation by a reflective meter (SmartProbe)
Basic metabolic panel | baseline and every 3 months
serum 1,25 dihydroxyvitamin D | baseline and 12 months
quality of life | baseline and 12 months
  questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: J C Gallagher, MD, Principal Investigator — Creighton University Medical Center
Locations (1):
- Creighton University Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gallagher JC, Kinyamu HK, Fowler SE, Dawson-Hughes B, Dalsky GP, Sherman SS. Calciotropic hormones and bone markers in the elderly. J Bone Miner Res. 1998 Mar;13(3):475-82. doi: 10.1359/jbmr.1998.13.3.475. PMID 9525348
- [Background] Holick MF, Siris ES, Binkley N, Beard MK, Khan A, Katzer JT, Petruschke RA, Chen E, de Papp AE. Prevalence of Vitamin D inadequacy among postmenopausal North American women receiving osteoporosis therapy. J Clin Endocrinol Metab. 2005 Jun;90(6):3215-24. doi: 10.1210/jc.2004-2364. Epub 2005 Mar 29. PMID 15797954
- [Background] Aloia JF, Talwar SA, Pollack S, Feuerman M, Yeh JK. Optimal vitamin D status and serum parathyroid hormone concentrations in African American women. Am J Clin Nutr. 2006 Sep;84(3):602-9. doi: 10.1093/ajcn/84.3.602. PMID 16960175
- [Derived] Smith LM, Gallagher JC. Effect of vitamin D supplementation on total and free 25 hydroxyvitamin D and parathyroid hormone. An analysis of two randomized controlled trials. J Intern Med. 2019 Dec;286(6):651-659. doi: 10.1111/joim.12950. Epub 2019 Jul 29. PMID 31215092
- [Derived] Smith LM, Gallagher JC, Kaufmann M, Jones G. Effect of increasing doses of vitamin D on bone mineral density and serum N-terminal telopeptide in elderly women: a randomized controlled trial. J Intern Med. 2018 Dec;284(6):685-693. doi: 10.1111/joim.12825. Epub 2018 Sep 17. PMID 30137647
- [Derived] Gallagher JC, Smith LM, Yalamanchili V. Incidence of hypercalciuria and hypercalcemia during vitamin D and calcium supplementation in older women. Menopause. 2014 Nov;21(11):1173-80. doi: 10.1097/GME.0000000000000270. PMID 24937025
- [Derived] Gallagher JC, Jindal PS, Smith LM. Vitamin D does not increase calcium absorption in young women: a randomized clinical trial. J Bone Miner Res. 2014;29(5):1081-7. doi: 10.1002/jbmr.2121. PMID 24166866
- [Derived] Gallagher JC, Peacock M, Yalamanchili V, Smith LM. Effects of vitamin D supplementation in older African American women. J Clin Endocrinol Metab. 2013 Mar;98(3):1137-46. doi: 10.1210/jc.2012-3106. Epub 2013 Feb 5. PMID 23386641
- [Derived] Gallagher JC, Sai A, Templin T 2nd, Smith L. Dose response to vitamin D supplementation in postmenopausal women: a randomized trial. Ann Intern Med. 2012 Mar 20;156(6):425-37. doi: 10.7326/0003-4819-156-6-201203200-00005. PMID 22431675